CLINICAL TRIAL: NCT03029858
Title: Programmed Death-ligand 1(PD-L1) and Other Immuno-markers Influenced by Osimertinib Treatment in Advanced Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: PD-L1 and Other Immuno-markers Influenced by Osimertinib Treatment in Advanced NSCLC Patients
Acronym: ATHENE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG1605; ESR-16-12177 (Other: Sponsor)
Record Dates: First submitted 2017-01-17; First posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Small Cell Lung Cancer, Polygonal Type
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tumor Formaldehyde Fixed-Paraffin Embedded (FFPE) tissue specimen collection • Tumor FFPE tissue specimen will be at least collected at baseline, disease progression and Response (optional) in sufficient amount (10 FFPE slices, thickness 4um, tumor cells≥25% and the area of necrotic tissues<10%).
  Blood specimen collection(optional)
  • The plasma specimen requirements for 10 ml blood will be collected at least at baseline, disease progression, and every 6 weeks, which is for detecting tumor mutation burden by QIAGEN Mix-561-Match Panel (561genes).
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No interventions will be taken in this Observational study — TAGRISSO(osimertinib/AZD9291）

SUMMARY:
The study will investigate whether PD-L1 and other immuno-markers will be influenced by osimertinib treatment in advanced epidermal growth factor receptor （EGFR）T790M positive advanced NSCLC patients. In addition, we will explore whether PD-L1 and other immuno-markers can predict the safety and efficacy of subsequent use of immune checkpoint inhibitors at the time of PD due to osimertinib resistance.

DETAILED DESCRIPTION:
Investigate whether PD-L1 and other immuno-markers will be influenced by osimertinib treatment in advanced EGFR T790M positive advanced NSCLC patients.

explore whether PD-L1 and other immuno-markers can predict the safety and efficacy of subsequent use of immune checkpoint inhibitors at the time of PD due to osimertinib resistance.

ELIGIBILITY:
Inclusion Criteria:

1. The patient enrolled in ASTRIS or patient who are eligible for the ASTRIS study.
2. The patient is willing to provide informed consent form to provide specimen before osimertinib treatment and at the time of PD.
3. Patients must be able to undergo a fresh tumor biopsy during screening or to provide an available tumor sample taken <2 months prior to screening.
4. Fine needle aspirate specimens are not acceptable.
5. Specimens from metastatic bone lesions are typically unacceptable unless there is confirmed soft tissue component.
6. The tumor specimen submitted to establish eligibility should be of sufficient quantity to allow for PD-L1 IHC and other biomarker analyses (if applicable) and is preferred in formalin-fixed paraffin embedded blocks.

Exclusion Criteria:

1. The patient does not have sufficient tumor tissue specimen available for detection.
2. The Patient who is unwilling to use the existing data from medical practice for scientific research.
3. The patient who received immunotherapy therapy before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) with locally advanced (stage IIIB) or metastatic (stage IV) NSCLC with confirmed T790M mutation, who have received prior EGFR-TKI therapy，These patients are those who were enrolled in ASTRIS（Real World Treatment Study of AZD9291 for Advanced/Metastatic EGFR T790M Mutation NSCLC） or patients who were eligible for the ASTRIS study.
  The study is a post observational study for ASTRIS study，and the patients would not take Osimertinib in this study any more.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2017-01; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Measure PD-L1 value | baseline and PD，up to 24 months
  Measure PD-L1 value Change by tumor cells（TC）/immune cells(IC) staining from the baseline to progressive disease（PD）
Measure PD-L1 expression positive rate (%) | baseline and PD，up to 24 months
  Measure PD-L1 expression positive rate (%) change from the baseline to progressive disease（PD）

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, M.D, Principal Investigator — Shanghai Chest hospital of Shanghai Jiaotong University
Locations (12):
- China (12):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Principal Cancer Hospital, Fuzhou, Fujian
  - The first Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The second affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital Oncology dept., Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital Respiratory dept., Shanghai, Shanghai Municipality
  - The first Affiliated hospital of Zhejiang University, Thoracic Oncology Dept., Hangzhou, Zhejiang
  - The first Affiliated hospital of Zhejiang University，Respiratory dept., Hangzhou, Zhejiang
  - The second Affiliated hospital of Zhejiang University of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Taizhou Hospital, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No